CLINICAL TRIAL: NCT01899391
Title: A Pilot Study of Gamma H2AX DNA Repair Foci Kinetics in Peripheral Blood Lymphocytes During Prostate Cancer Radiotherapy
Brief Title: Periperal Blood Lymphocytes During Prostate RT
Status: Withdrawn | Type: Observational
Why Stopped: Recuritment Challenges
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 09-0136-CE
Record Dates: First submitted 2013-06-11; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Right now it is not possible to predict which patients are going to react more to RT. Many things could affect patient's response to radiation. One of the factors is whether the person can repair damage to the genetic material (DNA/RNA) caused by the RT. There is some evidence that a certain protein called Gamma H2AX is involved in DNA damage and repair and this can be used to predict the sensitivity of individual patients. The investigators will be studying this protein: Gamma H2AX) in the blood samples of prostate cancer patients exposed to both computed tomography (CT) scan and RT treatment. This will help us to understand why different individuals show differences in side effects following RT.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate-risk prostate cancer patients (T1/T2N0M0 with either GS < 7 and PSA between 10-20 ng/ml or GS 7 and PSA less than 20 ng/ml).
* Planned for radical RT to the prostate with IMRT planning (79Gy/39fractions or 60 Gy/20 fractions).
* No contraindications to diagnostic CT scanning.
* Prostate volumes will be less than 80 cc to control the planning dose volume histogram (DVH) as much as possible in terms of rectal and bladder volumes.
* No known DNA repair disorders (e.g. family history of AT, BRCA1/2 or Li Fraumeni syndrome) or contraindications to radical pelvic RT.

Exclusion Criteria:

* Inability to provide informed consent.
* Patient having contraindications to diagnostic CT scan.
* Patients who have unobtainable data regarding previous therapy and their clinical outcome.
* Patients should not have any diagnostic X-rays or CAT scans 2 weeks prior to their enrollment into the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate-risk prostate cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Gamma H2AX in peripheral blood lymphocytes. | 1 year

SECONDARY OUTCOMES:
Gamma H2AX following RT planning (CT scan). | 1 year
Gamma H2AX during RT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bristow, MD, Principal Investigator — University Health Network, Princess Margaret Hospital